CLINICAL TRIAL: NCT05899634
Title: The Family Grocery Pilot: Examining the Use of Optimal Defaults in Online Grocery Shopping Among Families With 2-to-5-year-old Children.
Brief Title: The Family Grocery Pilot: Optimal Defaults in Online Grocery Shopping Among Families
Acronym: FGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Mackenzie J Ferrante, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00007317
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Obesity
Keywords: grocery shopping; online grocery shopping; obesity; behavioral economics; diet; children
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 - Recipes (No Intervention): Participants will receive healthy recipes (3 main meal + 1 snack/breakfast/lunch recipe per week of the two-week intervention).
- Group 2 - Default (Experimental): Participants will receive healthy recipes (3 main meal + 1 snack/breakfast/lunch recipe per week of the two-week intervention). In addition, in this group, participants' online grocery shopping carts will be pre-filled with ingredients corresponding to the provided recipes. They will be told that their cart has been filled with items that can be used to make recipes from the provided recipe cards, and that they can modify it as they like.
  Interventions: Behavioral: Defaults

INTERVENTIONS:
Behavioral: Defaults — Participants will receive healthy recipes (3 main meal + 1 snack/breakfast/lunch recipe per week of the two-week intervention). In addition, in this group, participants' online grocery shopping carts will be pre-filled with ingredients corresponding to the provided recipes. They will be told that their cart has been filled with items that can be used to make recipes from the provided recipe cards, and that they can modify it as they like.
  Arms: Group 2 - Default

SUMMARY:
The obesity epidemic continues to be a major public health concern, impacting nearly one-fifth of US children. One of the most robust predictors of childhood obesity risk is parental obesity and children who are overweight by age 5 are at increased risk for future obesity. A healthful diet is a significant part of preventing overweight and obesity and the home food environment can be a predictor of children's dietary intake. The goal of the proposed pilot study is to examine the feasibility and efficacy of a new family-based approach to early childhood obesity prevention, using optimal defaults in the form of pre-filled, default online grocery shopping carts to promote healthier grocery shopping among families with young children at risk for obesity, potentially influencing the home food environment and dietary intake.

DETAILED DESCRIPTION:
The goal of the proposed pilot study is to examine the feasibility and efficacy of a new family-based approach to early childhood obesity prevention, using optimal defaults in the form of pre-filled, default online grocery shopping carts to promote healthier grocery shopping among families with young children at risk for obesity. The specific aims are to: (1) test the feasibility and efficacy of a Defaults grocery shopping intervention designed to promote healthier grocery purchases among families with obesity, and (2) test effects of this intervention on the home food environment and dietary intake. To do this a randomized controlled intervention study has been designed, in which all study participants will receive 3 healthy recipes each week of a two-week intervention period, and intervention group will have their online grocery shopping carts pre-filled with corresponding ingredients.

Families who already grocery shop online and who have a 2-to-5-year-old child at home who is at increased obesity risk based on parental weight status will be randomly assigned to the intervention (Defaults) or control (Recipes) group. At baseline, all participants will complete a survey online and then will grocery shop as usual for two weeks. The baseline period will also serve as a run-in period, and participants who do not comply with study guidelines for baseline procedures will not be randomized for further participation. Participants will then be randomized and enter a two-week intervention period. During this period, all participants will be given recipe cards (3 main meal recipes + 1 snack/breakfast recipe each week), featuring healthful, budget friendly meals developed by dietitians. The Recipes group will continue to grocery shop as normal. The Defaults group will have their online shopping carts pre-filled with the study recipe ingredients. They will be told their cart has been filled with those items that could be used to make the healthful recipes on the recipe cards given to them. They may modify their carts as they choose. It is hypothesized that the Defaults group will have weekly grocery purchases with greater nutritional quality and lower energy content, compared to the Recipes group. It is hypothesized that the Defaults group will also have a home food environment with a greater nutritional quality score than the Recipes (via the Healthy Eating Index). Dietary intake of parents and children in the Defaults group will also have a higher nutritional quality, compared to the Recipes group, as indicated by food photography during 3 dinner meals during the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Participating parent/guardian must be at least 18 years old
* Must have a 2-to-5-year-old child in the household
* Must grocery shop online (via Instacart) from Tops, Wegmans, and/or Aldi stores at least 75% of the time
* Child must have at least one parent/guardian meeting criteria for overweight/obesity (BMI >25)
* Must speak English

Exclusion Criteria:

* Parent/guardian is under 18 years of age
* Does not have at least one 2-to-5-year-old child living in the household
* Does not shop online at Tops, Wegmans, and/or Aldi stores at least 75% of the time
* Child does not have at least one parent/guardian meeting criteria for overweight/obesity
* Does not speak English
* Has dietary restrictions or preferences that would not allow them to reasonably partake in the study (i.e., they would not be willing or able to buy/eat many of the staple foods included in default carts/recipe cards)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Nutritional Quality of Purchases in First Intervention Week | Intervention (Week 3)
  Receipt data from target grocery stores will be entered into nutrition software and used to quantify the number of foods purchased weekly for the household that correspond to Healthy Eating Index (HEI) food groups (e.g., fruits, dark green vegetables). These scores will be operationalized such that higher scores indicate more healthful food purchases aligning with HEI scoring.
Nutritional Quality of Purchases in Second Intervention Week | Intervention (Week 4)
  Receipt data from target grocery stores will be entered into nutrition software and used to quantify the number of foods purchased weekly for the household that correspond to HEI food groups (e.g., fruits, dark green vegetables). These scores will be operationalized such that higher scores indicate more healthful food purchases aligning with HEI scoring.
Change in Nutritional Quality of Purchases | Baseline (Weeks 1 and 2) and Intervention (Weeks 3 and 4)
  Receipt data from target grocery stores will be entered into nutrition software and used to quantify the number of foods purchased weekly for the household that correspond to HEI food groups (e.g., fruits, dark green vegetables). These scores will be operationalized such that higher scores indicate more healthful food purchases aligning with HEI scoring.
Energy Purchased in First Intervention Week | Intervention (Week 3)
  Receipt data from target grocery stores will be entered into nutrition software and used to calculate the total weekly calories purchased from target grocery stores.
Energy Purchased in Second Intervention Week | Intervention (Week 4)
  Receipt data from target grocery stores will be entered into nutrition software and used to calculate the total weekly calories purchased from target grocery stores.
Change in Energy Purchased | Baseline (Weeks 1 and 2) and Intervention (Weeks 3 and 4)
  Receipt data from target grocery stores will be entered into nutrition software and used to calculate the total weekly calories purchased from all grocery stores.
Cost of Groceries in First Intervention Week | Intervention (week 3)
  Total weekly dollars spent on grocery purchases from submitted receipts from target grocery stores
Cost of Groceries in Second Intervention Week | Intervention (week 4)
  Total weekly dollars spent on grocery purchases from submitted receipts from target grocery stores
Change in Cost of Groceries | Baseline (Weeks 1 and 2) and Intervention (Weeks 3 and 4)
  Total weekly dollars spent on grocery purchases from submitted receipts from target grocery stores

SECONDARY OUTCOMES:
Nutritional Quality of Home Food Environment | Intervention (Week 4)
  Data from a home food inventory will be used to create an HEI score based on the presence or absence of foods corresponding to HEI food groups (e.g., fruits, dark green vegetables). These scores will be operationalized such that higher scores indicate more healthful foods present in the home aligning with HEI scoring.
Meals and Meal Intake of Parent | Intervention (Week 4)
  Data from the food photographs will be used to create an HEI score based on the parent's consumption of foods (i.e., whether or not a food was consumed in any amount) which correspond to HEI food groups (e.g., fruits, dark green vegetables). These scores will be operationalized such that higher scores indicate more healthful foods present in the home aligning with HEI scoring.
Meals and Meal Intake of Child | Intervention (Week 4)
  Pre and post-meal photos with descriptions from children will be used to assess what foods are offered and quantify (1) if any of the foods were consumed and (2) the amount consumed (as a percentage) of individual foods offered during each of three dinner meals. Consumption of foods offered will be entered into nutrition software to calculate an estimate of calories consumed.
Nutritional Quality of Child's Intake | Intervention (Week 4)
  Data from the food photographs will be used to create an HEI score based on the child's consumption of foods (i.e., whether or not a food was consumed in any amount) which correspond to HEI food groups (e.g., fruits, dark green vegetables). These scores will be operationalized such that higher scores indicate more healthful foods present in the home aligning with HEI scoring.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Anzman-Frasca, PhD, Principal Investigator — University at Buffalo; Mackenzie J Ferrante, PhD, Principal Investigator — University at Buffalo
Locations (1):
- State University of New York at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anzman-Frasca S, Goldsmith J, Calabro A, Gambino K, Epstein LH, Leone LA, Wallenhorst B, Wilding GE, Ferrante MJ. Effects of an optimal defaults grocery shopping intervention on household grocery purchases of families with young children. Appetite. 2026 Mar 1;218:108397. doi: 10.1016/j.appet.2025.108397. Epub 2025 Nov 24. PMID 41297859